CLINICAL TRIAL: NCT05294159
Title: Implementing Long-Acting Novel Antiretrovirals - the ILANA Study
Brief Title: Implementing Long-Acting Novel Antiretrovirals
Acronym: ILANA
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IMP 218081
Record Dates: First submitted 2022-02-22; First posted 2022-03-24 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Human Immunodeficiency Viruses
Keywords: HIV-1; Long-acting antivirals; Implementation science
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinic-based PLH on CAB+RPV LA: All PWH participants will begin injections in the clinic setting in Phase 1. During Phase 1, PWH participants are screened and consented to participate in the study. During the screening phase, potential participants will be asked to identify their preferred location for phase 2 (decentralised site) and the reason for their preference. At the time of consent, patients will select their injection setting for Phase 2. Patients can select their preferred choice of setting until the 50 in-clinic numbers and 100 decentralised site places have been reached. After this, PWH participants will be allocated to the setting yet to reach its cap. In Phase 2, PWH participants will either continue to receive injection in clinic or receive injections from community nurses or clinic nurses at decentralised sites.
  Interventions: Other: The Feasibility of Intervention Measure (FIM) and Acceptability of Intervention Measure (AIM)
- Community-based PLH on CAB+RPV LA: All PWH participants will begin injections in the clinic setting in Phase 1. During Phase 1, PWH participants are screened and consented to participate in the study. During the screening phase, potential participants will be asked to identify their preferred location for phase 2 (decentralised site) and the reason for their preference. At the time of consent, patients will select their injection setting for Phase 2. Patients can select their preferred choice of setting until the 50 in-clinic numbers and 100 decentralised site places have been reached. After this, PWH participants will be allocated to the setting yet to reach its cap. In Phase 2, PWH participants will either continue to receive injection in clinic or receive injections from community nurses or clinic nurses at decentralised sites.
  Interventions: Other: The Feasibility of Intervention Measure (FIM) and Acceptability of Intervention Measure (AIM)

INTERVENTIONS:
Other: The Feasibility of Intervention Measure (FIM) and Acceptability of Intervention Measure (AIM) — The Feasibility and Acceptability of Intervention Measure (FIM and AIM) are used to evaluate the feasibilit and acceptability of our implementation strategies. The FIM and AIM is a validated implementation outcome measure where higher scores indicate greater feasibility and acceptability

SUMMARY:
This is a 12-month, dual arm, phase 4, open-label, multi-centre study examining the implementation of LA intra-muscular (IM) drugs in clinics and decentralised community-based settings in the UK.

DETAILED DESCRIPTION:
Cabotegravir and Rilpivirine (CAB+RPV) LA, is recommended in European US and British guidelines as a treatment for HIV-1 that allows PWH to receive a two-monthly injectable treatment, rather than daily pills. Providing injectable therapy in a system designed to provide and manage patients on oral treatments poses logistical challenges namely how resources are used to accommodate patient preference within a constrained health economy with capacity limitations. Exploring the use of alternative settings for injection, including community-based settings to deliver CAB+RPV LA, has the potential to expand options and potentially improve clinic capacity. Many PWH report high levels of stigma when attending the HIV clinic which can affect engagement with care, so receiving care in a community setting may provide additional choices and the possibility of receiving treatment in a less medicalized setting. Implementation studies in Europe are also assessing this in their countries.

The National Health Service (NHS) in the UK is a very specific health environment where people are entitled to treatment and care which is free at the point of delivery. Unlike other medical specialties where primary care physicians are responsible for prescribing treatment for chronic conditions, PWH are managed and receive their HIV treatment in HIV and sexual health clinics. For the circa 105K people with HIV in the UK, outcomes are excellent. More than 95% of those on treatment have undetectable viral loads. However, around 8100 people in the UK are not able to take oral ART successfully. US guidelines have specified that LA CAB+ RPV is particularly important for those who experience pill fatigue, stigma and have fears of inadvertent disclosure. This is highly relevant to the ethnically diverse population of people in the UK living with HIV, many of whom come from marginalized and minoritized communities in which stigma is rife and in whom the treatment outcomes are the poorest. Women, racially minoritized people and older people are chronically under-represented in HIV clinical trials which is why we have set recruitment caps to ensure we recruit 50% women, 50% ethnically diverse people and 30% over 50 years of age. This is to ensure that we go beyond lip-service and hold ourselves to account in designing our trials with peer researcher involvement from the outset and committing to include a more representative study population. We will achieve this by engaging actively with community organisations to ensure awareness of this implementation trials.

The study will be conducted at six large clinic sites both in London and outside of London. In this pragmatic real-world trial, each site will identify the most workable option to deliver of CAB+RPV LA according to SmPC license in the community setting within their region or borough.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Documented HIV-1 infection
* Virologically suppressed (HIV-1 RNA <50 copies/ml) on a stable antiretroviral regimen
* Able and willing to complete informed consent prior to inclusion
* No hepatitis B
* In accordance with EU license and NICE guidance

Exclusion Criteria:

* Based on contraindication for CAB LA, RPV LA, in accordance with EU license and NICE guidance
* Prior virologic failure on substances of NNRTI or INI class
* Resistance mutations to any substance of the NNRTI or INI class
* Prior exposure to CAB + RPV LA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 108 stable, virally suppressed PWH.
  To achieve representation of underrepresented groups in HIV studies, a cap will be set on recruitment of men at 50%, white participants at 50% and age under 50y at 70%.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Proportion of participants that agree or completely agree (average score of 4 or higher) on the Feasibility of Intervention Measure (FIM) (a validated method) | 12 months
  To evaluate feasibility of CAB and RPV LA administration at clinics in England and community based settings by patients

SECONDARY OUTCOMES:
Proportion of care provider and nurse participants that agree or completely agree (average score of 4 or higher) on the FIM and via qualitative interviews | At Day 0, 4 Months and 12 Months
  To evaluate feasibility of CAB and RPV LA administration at 6 English clinics and decentralised community settings by healthcare professionals (HCPs)
Proportion of care provider and nurse participants that agree or completely agree (average score of 4 or higher) Acceptability of Intervention Measure (AIM) (a validated method) | At Day 0, 4 Months and 12 Months
  To evaluate acceptability of CAB and RPV LA by participants and clinic staff
Proportion of community site representatives that agree or completely agree (average score of 4 or higher) score of on the FIM and AIM with in-depth qualitative interviews with community site representative | At 8 months and 12 months
  To evaluate feasibility and acceptability of CAB and RPV LA by community site representatives
Proportion of injections occurring within target window from target date (± 7 days of target date) | 12 months
  To describe adherence to dosing window by clinicians
Proportion of injections occurring after target window with/without use of oral ART | 12 months
  To describe adherence to dosing window by clinicians
Incidence and extent of oral bridging use | 12 months
  To describe adherence to dosing window by clinicians
Qualitative interviews with nurses to ascertain the utility of the Blueprints by Community Nurse or Clinic Nurse | 12 months
  To evaluate the utility of the Blueprints by Community Nurse or Clinic Nurse
Questionnaire checklist of Blueprint activities documentation to ascertain adaptations to Blueprints | 12 months
  To evaluate the fidelity to Blueprint by Community Nurse or Clinic Nurse
Qualitative interviews to ascertain the utility of Facilitation Calls to improve implementation from the HIV clinic staff, Community Nurses, Clinic Nurses | 12 months
  To evaluate the utility of Facilitation Calls to improve implementation from the HIV clinic staff, Community Nurses, Clinic Nurses
HIV Treatment Satisfaction Questionnaire (HIVTSQs-12) (a validated questionnaire) to assess and ascertain the change in treatment satisfaction score over time and by setting | 12 months
  To describe the change in treatment satisfaction score over time and by setting
Validated questionnaires to describe tolerability and acceptance of injections | 12 Months
  To describe tolerability and acceptance of injections
Validated questionnaires and qualitative interviews to ascertain participants' overall treatment experience preference and medical need for long-acting therapy | 12 Months
  To describe participants' overall treatment experience preference and medical need for long-acting therapy
Qualitative interviews to ascertain patient preference for setting they receive injections and the reasons for their choice | 12 Months
  To describe patient preference for setting they receive injections and the reasons for their choice

OTHER OUTCOMES:
Incidence of CAB and RPV LA related ADRs (adverse drug reactions) and all SAEs | 12 months
  To describe safety of CAB and RPV LA
Proportion of participants who do not progress to injections/discontinuation during oral lead in | 12 months
  To describe safety of CAB and RPV LA
Proportion of participants who discontinue CAB and RPV LA, for all cause, virological reasons or tolerability | 12 months
  To describe safety of CAB and RPV LA
Proportion of participants who are virologically suppressed (plasma HIV-1 RNA VL<50 c/mL) at month 4 and 12 (with +/- 6-week window) | 12 months
  To describe effectiveness of CAB and RPV LA
Proportion participants with VL ≥ 50 c/mL at M4 and M12 (with a +/- 6-week window | 12 months
  To describe effectiveness of CAB and RPV LA

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Orkin, Study Chair — QMUL
Locations (6):
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Royal Liverpool University Hospital, Liverpool
  - Blizard Institute, London
  - Royal Free Hospital NHS, London
  - Guys' and St Thomas' NHS Trust, London
  - Chelsea & Westminster NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Result] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Result] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Derived] Orkin C, Hayes R, Haviland J, Wong YL, Ring K, Apea V, Kasadha B, Clarke E, Byrne R, Fox J, Barber TJ, Clarke A, Paparini S. Perspectives of People With HIV on Implementing Long-acting Cabotegravir Plus Rilpivirine in Clinics and Community Settings in the United Kingdom: Results From the Antisexist, Antiracist, Antiageist Implementing Long-acting Novel Antiretrovirals Study. Clin Infect Dis. 2025 Jun 4;80(5):1103-1113. doi: 10.1093/cid/ciae523. PMID 39465685
- [Derived] Farooq HZ, Apea V, Kasadha B, Ullah S, Hilton-Smith G, Haley A, Scherzer J, Hand J, Paparini S, Phillips R, Orkin CM. Study protocol: the ILANA study - exploring optimal implementation strategies for long-acting antiretroviral therapy to ensure equity in clinical care and policy for women, racially minoritised people and older people living with HIV in the UK - a qualitative multiphase longitudinal study design. BMJ Open. 2023 Jul 9;13(7):e070666. doi: 10.1136/bmjopen-2022-070666. PMID 37423623